## Imperial College London



#### Al Clinician XP1 Informed Consent Form

Passive evaluation in operational environment of the Al Clinician decision support system for sepsis treatment

Version 1.1 – 6<sup>th</sup> January 2022

MAIN SPONSOR: Imperial College London

FUNDERS: NIHR/NHS-X

IRAS Project ID:297800 REC reference: 21/SC/0383 NCT number: NCT05287477

### Imperial College London

Research Governance and Integrity Team



#### **Informed Consent Form for Adults with Capacity**

Centre Number (if applicable): Study Protocol Number: EudraCT number (if applicable):

# INFORMED CONSENT FORM FOR SUBJECTS ABLE TO GIVE CONSENT

Full Title of Project: Passive evaluation in operational environment of the Al Clinician decision support system for sepsis treatment

Name of Principal Investigator: Professor Anthony Gordon Please initial box I confirm that I have read and understand the subject information sheet dated...... version ...... for the above study and have had the opportunity 1. to ask questions which have been answered fully. I understand that my participation is voluntary and I am free to withdraw at any time, 2. without giving any reason and without my medical care or legal rights being affected. I understand that sections of any of my research data may be looked at by responsible 3. individuals from Imperial College London, from NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to access my records that are relevant to this 4. research. I give/do not give (delete as applicable) consent for information collected about me to be 5. used to support other research in the future, including those outside of the UK. 6. I consent to take part in the above study. I give/do not give (delete as applicable) consent to being contacted to potentially taking 7. part in other research studies. Name of Subject Signature Date Name of Person taking consent Signature Date

1 copy for subject; 1 copy for Principal Investigator (ISF)